CLINICAL TRIAL: NCT03827954
Title: HeartMapp: A Closed-loop Assessment and Treatment Mobile Application for Heart Failure. A Pilot Clinical Trial
Brief Title: HeartMapp: Assessment and Treatment for Heart Failure
Acronym: HeartMapp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-1014-18; 1R43NR018415-01 (NIH)
Record Dates: First submitted 2019-01-23; First posted 2019-02-04 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure; Cognitive Impairment
Keywords: Heart failure; cognitive impairment; HeartMapp Mobile app; Self-care
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A single arm, open label, pilot clinical trial to examine feasibility and initial efficacy of the HeartMapp+CT (HeartMapp and computerized plasticity-based adaptive cognitive training).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): HeartMapp+CT
  Interventions: Other: HeartMapp+CT

INTERVENTIONS:
Other: HeartMapp+CT — HeartMapp+CT is a mobile system that includes physiological modules that support self-monitoring and exercises that promote heart health, and computerized plasticity-based adaptive cognitive training modules that train participants to enhance cognitive functions and ultimately heart failure outcomes.

SUMMARY:
In the current application, the investigators propose to elaborate upon, reconstruct and advance to pivotal trial readiness a recently validated mobile application (HeartMapp), designed for the ecological momentary assessment and treatment of individuals with Heart Failure (HF). Presently, HeartMapp includes physiological modules (PM) that support self-monitoring and exercises that promote heart health, and cognitive modules (CM) that track and enhance cognitive functions. During the first three-months, the investigators will finalize the cognitive training modules within HeartMapp and release through the quality management system. At the completion of software development, the investigators propose to test the relevant usage and progression variables of the algorithm that will be used to direct engagement with the app.

The investigators will conduct a single arm, open label, pilot clinical trial to examine feasibility and initial efficacy of the HeartMapp+CT (HeartMapp and computerized plasticity-based adaptive cognitive training). The term "CT" refers to computerized training. The study will enroll 32 adults aged 40 and older with a diagnosis of HF and over sample by 25% to reduce attrition for a total of 24 participants enrolled at the end. Participants will complete follow-up assessments at 3- and 6-months after enrollment.

DETAILED DESCRIPTION:
Heart failure (HF) is a progressive disease that affects 6.5 million Americans and is projected to reach 10 million by 2020. Presently, treatments for HF are largely comprised of drug therapies targeting pathophysiology and self-administered therapies that require patients to learn, accurately recall and routinely execute complex self-care practices. HF patients are expected to monitor their weight, diet and manage their medications, and are also required to recognize, monitor and report HF related symptoms. However, adopting self-care behaviors are often challenging for patients due to concomitant cognitive impairments, as shown in 30% to 80% of HF patients; a condition which is often complicated by insufficient social support. Multiple studies have shown a direct relationship between cognitive deficits and difficulty with self-care. Thus, there is currently an urgent unmet need for novel patient-centered interventions that are easy to use by older adults with HF that suffer cognitive difficulties and lack social support.

In the current application, investigators propose to elaborate upon, reconstruct and advance to pivotal trial readiness a recently validated mobile application (HeartMapp), designed for the ecological momentary assessment and treatment of individuals with HF. Presently, HeartMapp includes physiological modules (PM) that support self-monitoring and exercises that promote heart health, and cognitive modules (CM) that train participants to enhance cognitive functions. The Posit Science Corporation team of developer and neuroscientists will closely collaborate with investigators at University of South Florida (Drs. Athilingam and Labrador), inventors of the initial version of HeartMapp, to include a clinician-facing dashboard and reporting utility comprised of both PM and CM performance and progress tracking metrics. This Point-of-Care (POC) device will also aid clinical studies of cardiovascular, lung, and blood diseases and disorders by providing continuous monitoring data collected remotely to serve as an open channel between patients and clinicians. A recent usability study of the HeartMapp PM conducted by co-investigator Dr. Athilingam in 25 HF patients was successful; patients found the app easy to use, helpful and engaging. A concurrent pilot clinical trial that examined only CM in 17 HF patients demonstrated that CM improved memory, cognitive speed of processing, and showed trends for improved everyday function and HF self-care. Across all functional outcomes measured, the CM group showed better function post-training relative to controls. Similarly, in our prior research, and in the successful development of related products at Posit Science that demonstrated a core ability to develop multimodal (i.e., assessment and treatment) applications with compelling user experiences that drive strong performance improvements across multiple performance domains.

The investigators will conduct a single arm, open label, pilot clinical trial to examine feasibility and initial efficacy of the HeartMapp+CT (HeartMapp and computerized plasticity-based adaptive cognitive training). The study will enroll 32 adults aged 40 and older with a diagnosis of HF and over sample by 25% to reduce attrition for a total of 24 participants. Participants will complete follow-up assessments at 3- and 6-months after enrollment.

* The primary outcome is to test the feasibility and initial efficacy of using HeartMapp with computerized plasticity-based adaptive cognitive training (HeartMapp+CT), which will be quantified by measuring app usage and engagement with the apps. Engagement with cognitive training will be calculated as percentage of participants who complete 30 sessions of assigned cognitive training included in HeartMapp. App usability and engagement will be assessed by App access by participants; Accessing App components at least 80% of the days (72 days out of 90-days) will be used to determine app engagement.
* The secondary outcomes are improvement in cognitive function and HF self-care. If an effect sizes on Cohen's d of d=0.25 or greater relative to controls for these outcomes, HeartMapp will be considered potentially efficacious.
* Exploratory outcomes include improvement in quality of life, global health, medication adherence, heart rate variability and hospital admission. The investigators will calculate effect sizes using Cohen's d on these outcomes to inform future studies.

ELIGIBILITY:
Inclusion Criteria:

Selection of participants is based on their condition HF and is not based on gender or ethnic considerations, although these are expected to reflect the diverse population of the United States; ethnic minorities will be included when available and recruiting efforts will target a balanced enrollment.

* Age 40 years or above,
* Clinical diagnosis of HF as defined by the International Classification of Diseases (ICD-10 codes) and recent hospitalization for HF,
* New York Heart Association (NYHA) classification II-III,
* Ability to speak, understand and read English,
* Adequate hearing, as determined by response to a pure-tone stimulus at 70 decibels or better for 1 & 2 kHz in each ear, measured using the Welch-Allyn.
* Intact vision (visual acuity of 20/50 or better, as assessed by a Snellen chart per standard procedure).

Exclusion Criteria:

Participants meeting any of the following exclusion criteria at baseline will be excluded from study participation.

* Listed for heart transplant as status 1A,
* Enrolled in a palliative or hospice care program,
* Currently enrolled in another research study,
* Concurrent or previous participation in a cognitive training study within a month of the consent date,
* Self-reported vision, hearing, or motor difficulties that would interfere with the ability to complete the study interventions,
* Self-reported diagnosis of dementia, stroke, traumatic brain injury, brain tumor, or a neurological disorder that affects cognition or would interfere with the ability to benefit from the study intervention (e.g., Parkinson disease, multiple sclerosis), or any other unstable medical conditions that is predisposing to imminent cognitive or functional decline (e.g., undergoing chemotherapy or radiation),
* Presence of disability (e.g., aphasia) that may prevent them from completing study related activities,
* Severe depressive symptoms screened using PHQ-9 with score ≥16,
* History or current diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, delusion disorder, psychotic disorder, bipolar disorder, and/or mood congruent or mood incongruent psychotic features or disorders,
* Evidence of dementia with a score of <20 in the Montreal Cognitive Assessment, (MoCA),
* Shows signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs),
* Suicidal thoughts or ideations, or suicide-related behaviors using Columbia-Suicide Severity Rating Scale with 2 months of consent date.

Participants who are excluded due to depression, suicidal thoughts or ideation and/or dementia, poor vision or hearing will be referred to the appropriate professionals for thorough evaluation and treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Primary outcome (Feasibility of HeartMapp+CT app usage) | 3-months
  Above 80% usage of HeartMapp+CT will indicate feasibility of using the app.

SECONDARY OUTCOMES:
Cognitive outcomes (NIH-Examiner and Neuro QOL questionnaire) | up to 6-months (baseline and improvement at 3, and 6 months)
  Cognitive function will be measured using NIH-Examiner and Neuro QOL questionnaire provides a practical opportunity for multidimensional assessment in neurologic and cognitive assessment in clinical research or practice will be used. The internal consistency for this measure is (Cronbach alpha) of the 13 short forms ranged from 0.85 to 0.97. Higher scores on the cognitive measures will indicate improved cognition.
Heart failure Self-care (Self-Care of Heart Failure Index) | Up to 6-months (baseline and improvement at 3, and 6 months)
  Heart failure self-care will be assessed using the Self-Care of Heart Failure Index Cronbach's alpha of 0.81. The questionnaire measures three domains of self-care: Self-Care Maintenance, Self-management, and Self-Confidence. The questionnaire includes 15-items for a total score of 100. Lower scores indicates better self-care.
Quality of life related to Heart Failure (Kansas City Cardiomyopathy Questionnaire) | Up to 6-months (baseline and improvement at 3, and 6 months)
  Quality of life will be measured using Kansas City Cardiomyopathy Questionnaire that include five clinically relevant domains: physical limitations, HF symptom (frequency, severity, and change over time), quality of life, social interference, and self-efficacy. (Cronbach's alpha of 0.66-0.95) higher composite scores indicate better quality of life.
Physical and Mental Health (PROMISE short-form scale) | Up to 6-months (baseline and improvement at and 6 months)
  Global physical and mental health will be measured using the PROMISE short-form scale that measures (4 items on overall physical health, physical function, pain, and fatigue) and global mental health (4 items on quality of life, mental health, satisfaction with social activities, and emotional problems) with internal consistency .81-.86, respectively. Lower score of both domains indicates better physical and mental health.
Clinical outcomes (6-minute Walk Test) | Up to 6-months (baseline and improvement at 3, and 6 months)
  Physical capacity will be measured by distance walked using 6-minute Walk Test
Heart rate Variability | Up to 6-months (baseline and improvement at 3, and 6 months)
  Heart rate variability measured using BioPatch to determine improvement overtime

OTHER OUTCOMES:
Exploratory outcomes (number of hospital and er admissions) | Up to 6-months (decreased at 3, and 6 months)
  Number of hospital admissions and emergency room admissions

CONTACTS AND LOCATIONS:
Overall Officials: Ponrathi R Athilingam, PhD, Principal Investigator — University of South Florida; Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data of participants collected via REDCap will be made available to an unblinded research staff at Posit Science Corporation, San Francisco, CA, However, the PI to whom the grant is awarded will only have access to de-identified data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code